CLINICAL TRIAL: NCT03895580
Title: Supermarket and Web-Based Intervention Targeting Nutrition (SuperWIN) for Cardiovascular Risk Reduction
Acronym: SuperWIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: The Kroger Company (Unknown); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Dylan Steen, Director of Clinical Trials and Population Health Research, UC Heart, Lung, and Vascular Institute, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20168163
Record Dates: First submitted 2019-03-21; First posted 2019-03-29 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Obesity; Hypertension; Hyperlipidemias; Diet Modification
MeSH Terms: conditions — Obesity; Hypertension; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Due to COVID-19, recruitment and all in-person visits had to be temporarily stopped due to safety concerns in March 2020. Due to this stoppage, 20 randomized subjects could not complete their in-person study visits or data collection as per protocol. These 20 subjects will be excluded from all primary analyses, including the primary endpoint. Recruitment and in-person visits resumed in June 2020. To account for the exclusion of these 20 subjects, we randomized 267 subjects by the end of the study in order to have 247 subjects available for the primary analyses (e.g. 267-20= 247). A prespecified COVID impact analysis has been included in the statistical analysis plan.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (No Intervention): Medical nutrition therapy session with no further dietary counseling throughout the study.
- Group 2 (Experimental): Medical nutrition therapy session plus in-store point-of-purchase (POP) education.
  Interventions: Other: In-store POP education
- Group 3 (Experimental): Medical nutrition therapy session plus combined in-store/online point-of-purchase (POP) education.
  Interventions: Other: In-store POP education; Other: Online POP education

INTERVENTIONS:
Other: In-store POP education — Six in-store nutrition counseling sessions with a registered dietitian nutritionist.
  Arms: Group 2; Group 3
Other: Online POP education — Education on the use of an online grocery shopping, an online recipe tool, a grocery pickup service, a home grocery delivery service, and a phone application that promotes healthy food selection.
  Arms: Group 3

SUMMARY:
The Supermarket and Web-based Intervention targeting Nutrition (SuperWIN) for cardiovascular risk reduction is a novel, randomized controlled trial aimed at increasing diet quality and decreasing cardiovascular risk. SuperWIN will deliver individualized, nutrition education at the point-of-purchase (POP), either in the aisles of the physical store or via online shopping platforms coupled with other modern software tools.

DETAILED DESCRIPTION:
This study is designed to test whether individualized, POP nutrition education can improve dietary quality. The two interventions to be evaluated in SuperWIN will utilize either an in-store POP education strategy or a combined online/in-store POP education strategy in participants with at least one cardiovascular disease risk factor. The POP education interventions will be enhanced with sophisticated, provider- and participant-facing, food-purchasing metrics, a novel counseling tool that here-to-fore has not been studied in regard to changing food shopping behavior. The primary outcome measure is the Dietary Approaches to Stop Hypertension (DASH) score, a measure of adherence to the DASH dietary pattern. The study is well-powered to test at Day 90: 1) whether any POP education intervention strategy (both intervention arms pooled) improves the DASH score compared to the control arm and 2) whether an improvement in DASH score depends on the POP education strategy utilized.

Both POP education strategies will be delivered within a supermarket-based retail clinic and will utilize the aisles and products of the supermarket. The interventions will be delivered by a registered dietitian nutritionist (RDN). The online portion of the combined online/in-store education POP strategy will include online grocery shopping, online recipe resources, a grocery pickup or home delivery service, and a phone application to better select healthy foods.

Both strategies will be offered in addition to a "standard of care" medical nutrition therapy session. The DASH dietary pattern has been empirically tested and shown to favorably modify blood pressure, blood cholesterol, insulin sensitivity, and weight status.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 to ≤75 years on the start date of the study (Day 0)
2. Speak, write, read English fluently
3. In-person outpatient visit with a UC Health primary care network (PCN) provider within the last 12 months
4. Major food planner of their household, which may include planning, purchasing, and/or preparing greater than 50% of the meals or foods consumed at home
5. Existing shopper at a study site Kroger (≥50% of grocery store food dollars spent at Kroger) with a Kroger Loyalty ID number
6. Willing to use a new individual Kroger Loyalty ID number for the duration of the study
7. Access to a home desktop or laptop computer with reliable internet access
8. Access to an email account that can be used for the duration of the study
9. Able to independently purchase and prepare food:

   1. Reliable transportation to participating Kroger store
   2. Ability to stand for significant periods of time to grocery shop and prepare food at home
   3. Tools and equipment needed to prepare own food at home, such as a kitchen equipped with basic cooking tools (e.g. burner, pan, spatula, sink)
10. Presence of a cardiovascular risk factor(s) (at least one):

    1. Hypertension (defined by one of the following):

       * Blood pressure measurement: systolic blood pressure (SBP) 130-189 mm Hg and/or diastolic blood pressure (DBP) 80-109 mm Hg (at Visit #1)
       * Current treatment with an oral medication prescribed by a physician for blood pressure lowering (defined by one of the following):

         1. Beta blockers
         2. Diuretics (e.g. thiazide or thiazide-like diuretics, loop diuretics, aldosterone antagonists, potassium-sparing diuretics)
         3. Angiotensin-converting enzyme inhibitors
         4. Angiotensin II receptor blockers
         5. Direct renin inhibitors (i.e. aliskiren)
         6. Calcium channel blockers (dihydropyridine and nondihydropyridine)
         7. Calcium alpha2-agonist and other centrally acting drugs (e.g. clonidine)
         8. Direct vasodilators (e.g. hydralazine)
    2. Body-mass index (BMI) measurement ≥30 kg/m2 (at Visit #1)
    3. Hypercholesterolemia (defined by one of the following):

       * Low density lipoprotein cholesterol (LDL-C) 130-189 mg/dl (at Visit #1)
       * Current treatment with a medication prescribed by a physician for hypercholesterolemia (defined by one of the following):

         1. Statins
         2. Proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors
         3. Absorption inhibitors (i.e. ezetimibe)
         4. Fibrates
         5. High-dose niacin (≥1 g per day)
         6. Bile acid sequestrants (e.g. cholestyramine)

Exclusion Criteria:

1. Unwillingness or inability to modify current diet
2. Actively engaged in another dietary intervention or taking a weight-loss supplement
3. SBP ≥190 mm Hg or DBP ≥110 mm Hg (at Visit #1)
4. Low-density lipoprotein cholesterol (LDL-C) ≥190 mg/dl, triglycerides (TG) ≥600 mg/dl, or glucose ≥400 mg/dl (at Visit #1)
5. Evidence of prior diagnosis of severe chronic kidney disease (CKD) defined by electronic health record codes for dialysis, CKD Stage 4 or 5 and/or last estimated glomerular filtration rate (eGFR) ≤30 ml/min/1.732 [based on Modification of Diet in Renal Disease (MDRD) formula]
6. Active cancer other than non-melanoma skin cancers (i.e. basal cell carcinoma or squamous cell carcinoma)
7. Diagnosis of celiac disease, ulcerative colitis, or Crohn's disease
8. High risk for alcohol use disorder:

   1. ≥21 drinks a week (men)
   2. ≥14 drinks a week (women)
9. Women who are pregnant or plan to become pregnant within the next 6 months from the start of the study (Day 0)
10. Food allergies requiring a specialized diet, including allergies to dairy products, eggs, peanuts, tree nuts, soy, gluten-containing wheat and grains, fish, and shellfish
11. Previous visit at TLC for diet counseling
12. Previous use of the Kroger's online shopping platform (Kroger.com or the Kroger app)
13. Participant lives greater than 20 miles from any participating Kroger study store (defined by zip codes)
14. Women, Infants, and Children (WIC) beneficiaries in their household

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Dietary Approaches to Stop Hypertension (DASH) score | Baseline with follow-up measures at 90 days and 180 days. Primary tests are between baseline and 90 day timepoint.
  The DASH score will be calculated from food group analyses obtained from means of three 24-hour dietary intake recalls at each time-point. This DASH score is a 90-point continuous score used to measure change in overall dietary quality in response to an intervention. Given that the dietary focus of the SuperWIN interventions is the DASH dietary pattern, the DASH score will be used as a measure of adherence to a DASH eating pattern. Higher values indicate greater adherence.

SECONDARY OUTCOMES:
Change in systolic arterial blood pressure | Baseline with follow-up measures at 90 days and 180 days.
  Measured in the arm. Units: mm Hg
Change in diastolic arterial blood pressure | Baseline with follow-up measures at 90 days and 180 days.
  Measured in the arm. Units: mm Hg
Change in body mass index | Baseline with follow-up measures at 90 days and 180 days.
  Height and weight measured. Units: kg/m2
Change in non-high density lipoprotein cholesterol (Non-HDL-C) | Baseline with follow-up measures at 90 days and 180 days.
  Total cholesterol minus HDL-C. Units: mg/dL
Change in total cholesterol | Baseline with follow-up measures at 90 days and 180 days.
  Measured. Units: mg/dL
Change in triglycerides | Baseline with follow-up measures at 90 days and 180 days.
  Measured. Units: mg/dL

OTHER OUTCOMES:
Change in waist circumference | Baseline with follow-up measures at 90 days and 180 days.
  Measured. Units: cm
Change in food literacy | Baseline with reassessment at 90 days.
  Assessed by participant survey.
Participant experience and feedback | Collected at 90 days.
  Assessed by participant survey.
Dietitian experience and feedback | Collected at 90 days.
  Assessed by dietitian survey.

CONTACTS AND LOCATIONS:
Overall Officials: Dylan L Steen, MD, MS, Principal Investigator — University of Cincinnati; Sarah C Couch, RD, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center - UC Health, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steen DL, Helsley RN, Bhatt DL, King EC, Summer SS, Fenchel M, Saelens BE, Eckman MH, Couch SC. Efficacy of supermarket and web-based interventions for improving dietary quality: a randomized, controlled trial. Nat Med. 2022 Dec;28(12):2530-2536. doi: 10.1038/s41591-022-02077-7. Epub 2022 Dec 1. PMID 36456831